CLINICAL TRIAL: NCT01102517
Title: A Trial on Video-assisted Thoracoscopic Surgery and Axillary Thoracotomy for Resection of Early-stage Non-small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shanghai Chest Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); Shenzhen People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Long, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007039
Record Dates: First submitted 2010-04-06; First posted 2010-04-13 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Clinical; Early-stage
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VATS group (Experimental): video-assisted thoracoscopic surgery
  Interventions: Procedure: video-assisted thoracoscopic surgery
- axillary thoracotomy (Other): Control group
  Interventions: Procedure: axillary thoracotomy

INTERVENTIONS:
Procedure: video-assisted thoracoscopic surgery — video-assisted thoracoscopic surgery
  Arms: VATS group
Procedure: axillary thoracotomy — axillary thoracotomy lobectomy
  Arms: axillary thoracotomy

SUMMARY:
The purpose of this study is to establish the effects of VATS lobectomy for early-stage non-small cell lung cancer.

The aims of this study are:

1. To evaluate the early clinical benefits of VATS lobectomy when compared with the axillary thoracotomy.
2. To evaluate the late effects of VATS lobectomy on survival and quality of life when compared with axillary thoracotomy.
3. To establish the normative pattern of VATS lobectomy for early-stage non-small cell lung cancer.
4. To explore the indication of VATS lobectomy for the lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Early stage NSCLC and no metastasis of hilum of lung and mediastinum lymph nodes (short diameter ≤ 1 cm) on computed tomography (CT) scan;
* No medical contraindications to lung resection
* Age ≤ 75 years old and ≥18 years old;
* Sign the informed consent form.

Exclusion Criteria:

* Evidence of invasion into neighboring organs;
* Extensive pleura adhesion;
* Central lesion;
* Not suitable for single-lung ventilation;
* Had history of thoracotomy and radiation for thoracic region ;
* Pregnancy or lactation female patients;
* Cannot sign the informed consent form because of psychological, family and society factors;
* Had history of other malignant tumors within 5 years except for non-melanoma cutaneous cancer, uterine cervix cancer in situ and curative early-stage carcinoma of prostate;
* Participants can not accept operation for other uncontrolled factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2010-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival and overall survival | 5 years

SECONDARY OUTCOMES:
Quality of life | the first year after the surgery
  Lung Cancer Symptom Scale
Postoperative pulmonary function | the first three months after the surgery
Postoperative Karnofsky performance status | the first year after the surgery
Postoperative Chest Pain | the first year after the surgery
  visual analogue scale and Wong-Baker FACES Pain Rating Scale
Perioperation data | perioperation
  operation time, intraoperative blood loss, chest tube drainage amount, duration of the chest tube placement, and duratio
Cytokines response | the first 48 hours after the surgery
  IL-2,IL-4,IL-6,IL-10,TNF,IFN-r

CONTACTS AND LOCATIONS:
Overall Officials: Hao Long, professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] 1.Bethencourt DM, Holmes EC. Muscle-sparing posterolateral thoracotomy. Ann Thorac Surg. 1988;45(3):337-339. 2.Ginsberg RJ. Alternative (muscle-sparing) incisions in thoracic surgery. Ann Thorac Surg. 1993;56(3):752-754. 3.Weissberg D, Kaufman M. Technical aids in surgery. Two muscle-sparing thoracotomies--techniques and indications. S Afr J Surg. 1990;28(1):17-19. 4.Akçali Y, Demir H, Tezcan B. The effect of standard posterolateral versus muscle-sparing thoracotomy on multiple parameters. Ann Thorac Surg. 2003;76(4):1050-1054. 5.Hazelrigg SR, Landreneau RJ, Boley TM, et al. The effect of muscle-sparing versus standard posterolateral thoracotomy on pulmonary function, muscle strength, and postoperative pain. J Thorac Cardiovasc Surg. 1991;101(3):394-400. 6.Kutlu CA, Akin H, Olcmen A, et al. Shoulder-girdle strength after standard and lateral muscle-sparing thoracotomy. Thorac Cardiovasc Surg. 2001;49(2):112-114. 7.Khan IH, McManus KG, McCraith A, et al. Muscle sparing thoracotomy: a biomechanical analysis confirms preservation of muscle strength but no improvement in wound discomfort. Eur J Cardiothorac Surg. 2000;18(6):656-661. 8.Baeza OR, Foster ED. Vertical axillary thoracotomy: a functional and cosmetically appealing incision. Ann Thorac Surg. 1976;22(3):287-288.
- [Derived] Long H, Tan Q, Luo Q, Wang Z, Jiang G, Situ D, Lin Y, Su X, Liu Q, Rong T. Thoracoscopic Surgery Versus Thoracotomy for Lung Cancer: Short-Term Outcomes of a Randomized Trial. Ann Thorac Surg. 2018 Feb;105(2):386-392. doi: 10.1016/j.athoracsur.2017.08.045. Epub 2017 Dec 2. PMID 29198623